CLINICAL TRIAL: NCT06980987
Title: Pain Prevalence and Management in Neurological and Neurosurgical in Patients- the PAINN Study
Brief Title: The PAINN Study - a Pilot Cross Sectional Study
Acronym: PAINN
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Suzanne Forsyth Herling, Associate professor, RN, Rigshospitalet, Denmark
Other Study IDs: P-2023-98; Rigshospitalet (Other: Neurocentret)
Record Dates: First submitted 2025-05-12; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Hospitalized Patient; Home Mechanical Ventilation; Pain; Pain Management
Keywords: Pilot cross sectional study; Neurological patients; Home mechanical ventilation
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pain prevalence in hospitalized patients has been reported between 65% and 75%, indicating poor and/or insufficient management. In addition, pain prevalence has been estimated for separate groups of individuals with specific neurological/neurosurgical conditions (25% - 84%) and the overall prevalence was calculated as 36% (95% CI: 31% - 42%). However, investigations on prevalence of pain in Danish neurologic inpatients is scarce, which may indicate an overlooked symptom in local neurologic settings.

This project was a cross-sectional investigation to identify pain prevalence, intensity and interference in admitted patients needing home menicahal ventilation (HMV) and we conducted as an exploratory investigation to collect data from the patients by pain questionnaires/instruments, observation of patients' pain behavior and physiologic parameters. The main patients' diagnoses were spinal cord injury, amyotrophic lateral sclerosis, cerebral palsy, spinal muscular atrophy, and defects from birth such as tracheomalacia. The study included 40 participants, all recruited from Respiratory Center East, University of Copenhagen, Rigshospitalet

ELIGIBILITY:
Inclusion Criteria: persons hospital admitted, minimum 18 years old, provided informed consent (provided by the patient or patient's relative).

Exclusion Criteria: persons who did not understand written and spoken Danish or denied participating in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospital admitted patients, needing home mechanical ventilation for neurological disease or trauma,
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-01-03 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Brief Pain Inventory | 24 hours
  Pain impact on domains of every day life.

SECONDARY OUTCOMES:
GAD-7 | 24 hours
  Anxiety/depression
PHQ-9 | 24 hours
  Anxiety/depression
The Barthel Index | 24 hours
  Physical performance status

CONTACTS AND LOCATIONS:
Locations (1):
- Respirations center east, Copenhagen, Ø, Denmark

IPD SHARING:
Plan to Share IPD: No
It is a quality assurance pilot project.